CLINICAL TRIAL: NCT02860923
Title: Multicentre Double-blind Randomized Clinical Trial Assessing Efficacy and Safety of Exenatide in the Treatment of Hypothalamic Obesity After Craniopharyngioma Therapy
Brief Title: Efficacy and Safety of Exenatide in the Treatment of Hypothalamic Obesity After Craniopharyngioma Therapy
Acronym: CRANIOEXE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHUBX 2012/17
Record Dates: First submitted 2016-06-24; First posted 2016-08-09 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Craniopharyngiomas; Hypothalamic Obesity
Keywords: glucagon-like peptide-1; exenatide; placebo; multicenter trial
MeSH Terms: conditions — Craniopharyngioma; Sexual Infantilism | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide (Experimental): Treatment with exenatide at the initial dose of 5 µg x 2/day (subcutaneously administered) during 4 weeks, and treatment with 10 µg x 2/day during 5 months.
  Interventions: Drug: Exenatide
- Placebo (Placebo Comparator): Patients will be maintained on placebo (injected subcutaneously, twice a day) with the same dose and frequency than exenatide arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exenatide
  Arms: Exenatide
Drug: Placebo
  Arms: Placebo

SUMMARY:
This hypothalamic obesity is associated with serious metabolic and psychosocial consequences.

The purpose of the study is to compare the change of body weight after 6 months treatment with a lifestyle intervention + exenatide compare to the one after the same lifestyle intervention+ placebo in adults patients suffering from a hypothalamic obesity due to treatment of craniopharyngioma.

DETAILED DESCRIPTION:
The development of glucagon-like peptide-1 (GLP-1) analogues might be a solution since native GLP-1 suppresses appetite and energy intake in both normal weight and obese individuals as well as in people with type 2 diabetes and delays gastric emptying. The underlying mechanisms that mediate the effects of weight involve not only central regions like the hypothalamus and the solitary tractus nucleus and area postrema but also peripheral regions as the gastrointestinal tract. These extra hypothalamic effects are of particular interest in the cases of obesity due to hypothalamic lesions.

Exenatide is a glucagon-like peptide-1 (GLP-1) analogue with a high structural homology to human GLP-1, a gut derived incretin hormone. Since exenatide causes a dose-dependent weight loss, decreasing concentration of glycosylated haemoglobin as well as improving ß-cell function and systolic blood pressure, it could be an attractive treatment for both type 2 diabetes and obesity. In a double-blind placebo-controlled 24-week trial, it has been recently shown that non diabetic obese patients maintained on exenatide 10µg x 2/j lost significantly more weight than did those on placebo (5.1 kg versus 1.6).

ELIGIBILITY:
Inclusion Criteria:

* They are between 18 and 75 yrs.
* They had been diagnosed with a craniopharyngioma treated by surgery and/or irradiation without sign of recurrence.
* They have a BMI upper than 30kg/m² with intractable weight gain following therapy for craniopharyngioma.
* They demonstrate at least one other endocrinopathy, as a marker of hypothalamic damage.
* All pituitary deficiencies are correctly treated.
* They gave their written, informed consent before the beginning of the study.

Exclusion Criteria:

* They have type 1 diabetes.
* They have type 2 diabetes treated with insulin.
* Acidocetosis.
* Bariatric surgery
* Previous personal history of thyroid or pancreatic cancer.
* Hypercalcitoninemia.
* They have been previously treated by GLP1 analogs.
* Hypertriglyceridemia upper than 5g/l
* They had previously demonstrated voluntary weight loss during the three previous months.
* They are under the age of 18 years or over the age of 65 yrs.
* They are maintained on medical treatment against obesity.
* They are receiving supraphysiologic hydrocortisone therapy (upper than 30 mg/jour).
* Their GH status change during the course of the study.
* Exenatide is contraindicated.
* Psychological and/or medical problems that would create difficulties for the patient to comply with the study protocol are present.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Compare body weight change thanks to weighing machine | baseline and 6 months
  The primary outcome will be assessed by a weighing machine that measure until 200 kg.

SECONDARY OUTCOMES:
Treatment tolerance thanks to digestive parameters | 6 months
  Tolerance will be assessed by the presence of:
  - Nauseas, vomiting.
Treatment tolerance thanks to dermatologic parameter | 6 months
  Tolerance will be assessed by the presence of:
  - Injection-site symptoms.
Treatment tolerance thanks to pulse rate | 6 months
  Tolerance will be assessed by the presence of :
  - Increasing of pulse rate.
Treatment tolerance thanks to Beck scale | 6 months
  Tolerance will be assessed by the presence of :
  - Anxiety by Beck scale.
Treatment tolerance thanks to HAD scale | 6 months
  Tolerance will be assessed by the presence of :
  - depression evaluated by HAD scale.
Treatment tolerance thanks to enzymatic parameters | 6 months
  Tolerance will be assessed by the presence of :
  - Increasing of pancreatic enzymes.
Treatment tolerance thanks to glycemia parameter | 6 months
  Tolerance will be assessed by the presence of :
  - Hypoglycaemia
Assess cardiovascular risks thanks to glucose profil | 6 months
  Levels of blood glucose and insulin, oral glucose tolerance testing, haemoglobin A1C
Assess cardiovascular risks thanks to lipid profil | 6 months
  Levels of HDL cholesterol, triglycerides, LDL cholesterol.
Assess cardiovascular risks thanks to metabolic parameters | 6 months
  The metabolic parameters considered:
  - Body composition (Dual energy-ray absorptiometry) and abdominal obesity (waist circumference).
Assess eating behaviour thanks to physiological parameters | 6 months
  The eating behaviour will be evaluated by:
  - Plasma level of ghrelin measured after an overnight fast.
Assess eating behaviour thanks to energy intake | 6 months
Assess eating behaviour thanks to Three factor eating | 6 months
  The eating behaviour will be evaluated by:
  - Scores of restriction, hunger and disinhibition (French version of the Three factor Eating Questionnaire).
Assess eating behaviour thanks to visual analogic scales | 6 months
  The eating behaviour will be evaluated by:
  - Scores of desire to eat, hunger and fullness at visual analogic scales.
Assess quality of life thanks to Beck questionnaire | 6 months
  The quality of life will be assessed by:
  - Scores of depression (short questionnaire of Beck).
Assess quality of life thanks to ORWELL questionnaire | 6 months
  The quality of life will be assessed by:
  - Scores of quality of life (ORWELL questionnaire).
Assess energy expenditure thanks to physical activity | 6 months
  The energy expenditure will be estimated thanks to pedometer.
  - Resting metabolic rate (indirect calorimetry).
Assess energy expenditure thanks to indirect calorimetry | 6 months
  The energy expenditure will be estimated thanks to:
  - Resting metabolic rate

CONTACTS AND LOCATIONS:
Overall Officials: Paul Perez, Dr, Study Chair — University Hospital, Bordeaux; Blandine Gatta-Cherifi, Pr, Principal Investigator — University Hospital, Bordeaux
Locations (11):
- France (11):
  - CHU d'Angers, Angers
  - CHU de Brest, Brest
  - CHU de Grenoble, Grenoble
  - CHU de Lyon, Lyon
  - APHM, Marseille
  - Hôpital Bicêtre, Paris
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Pitié Salpétrière (APHP), Paris
  - Hôpital Haut-Lévêque, Pessac
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No